CLINICAL TRIAL: NCT02081742
Title: COMPARATIVE STUDY OF THE EFFICACY OF TWO NON-INVASIVE IMAGING TECHNIQUES IN POPULATION SCREENING FOR COLORECTAL CANCER (CRC): COLON CAPSULE AND VIRTUAL COLONOSCOPY
Brief Title: Comparative Study of Colon Capsule and Virtual Colonoscopy (VICOCA)
Acronym: VICOCA
Status: Completed | Type: Observational
Sponsor: Begoña González Suárez (Other)
Collaborators: Norgine (Industry); Medtronic - MITG (Industry)
Responsible Party: Sponsor-Investigator, Begoña González Suárez, MD PhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Other Study IDs: CCV-003
Record Dates: First submitted 2013-09-16; First posted 2014-03-07 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Colonic Polyps; Adenoma
Keywords: Colonoscopy, CT colonography, Colon capsule
MeSH Terms: conditions — Colonic Polyps; Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Summary Colorectal cancer (CRC) represents the second leading cause of cancer deaths in Spain (11,000 deaths per year). Screening of the population over 50 years of age with no significant history (intermediate risk) is recommended, but which screening method is best for promoting adherence in this type of patient has not been well established. There are currently two screening methods that are less invasive than conventional colonoscopy and seem to have higher sensitivity than the test for faecal occult blood (FOBT). These two methods are the colon capsule, which consists in ingesting a capsule that takes photographs of the colon, and virtual colonoscopy, which is a radiological technique.

Objectives: 1. To demonstrate that virtual colonoscopy and colon capsule are effective CRC screening techniques in the intermediate risk population, with diagnostic rates comparable to conventional colonoscopy (concordance). 2. To compare the diagnostic rates of the colon capsule and virtual colonoscopy with respect to the size and characteristics of the lesions visualised. 3. To compare the participation rates for each screening strategy and identify the factors that influence participation (individual, family, and socioeconomic factors as well as those relating to the doctor).

DETAILED DESCRIPTION:
Based on the fact that CRC is an important healthcare issue and that there is enough evidence to show that this disease, if diagnosed early, is curable and at a reasonable cost, the European Community Council, in 2003, issued directives that member states would make population screening for CRC a priority in their healthcare planning. Thus, Spain's Ministry of Health and Consumer Affairs included population screening for CRC in its National Healthcare Plan as a priority action within the Comprehensive Plan against Cancer (PICA), which was required to be implemented by the year 2007.

The screening tools we currently have are not ideal either because, like the test for faecal occult blood (FOBT), which is the most evaluated to date, they are not sensitive enough or, like conventional colonoscopy, they are not risk-free. All of this means that population adherence is limited.

In this study, we wish to compare two new diagnostic techniques for CRC (colon capsule and virtual colonoscopy) that, although recently introduced into the healthcare system, have sufficient scientific evidence to confirm that they are effective and possibly cost-effective techniques.

The population we are concerned with in this study is the healthy population-men and women 50-69 years of age with no significant history. Therefore, the screening method we offer must be the least invasive and the most comfortable method possible so that good compliance is achieved. This means techniques that are painless and essentially harmless in comparison with conventional colonoscopy. If we were to observe higher concordance between these techniques and conventional colonoscopy in terms of detecting lesions, we would use the latter strictly for therapeutic reasons in this population, thereby significantly reducing the complications associated with it.

Objectives

Main objectives:

1. To demonstrate that virtual colonoscopy and colon capsule are effective CRC screening techniques in the intermediate risk population, with adenoma diagnostic rates comparable to conventional colonoscopy.
2. To compare the diagnostic capabilities of the colon capsule and virtual colonoscopy with those of conventional colonoscopy with respect to the size and characteristics of the lesions (especially lesions that are flat or smaller than 6 mm).
3. To analyse the population's participation rate for each screening strategy and identify the factors that influence participation (individual, family, and socioeconomic factors as well as those relating to the doctor or the diagnostic procedure).

Secondary objectives:

1. To evaluate the rate of minor and major complications for each screening strategy.
2. To analyse the rate of false positives and false negatives for the colon capsule and virtual colonoscopy in comparison with conventional colonoscopy.

Methodology Type of study Randomised, and controlled study.

Study subjects

Inclusion Criteria:

The main objective in this study is compare two non-invasive techniques in the study of colorectal cancer. When we calculate the sample size we observed that we need more than 1000 patients per group. In this moment this study is very expensive and it is not feasible. Our proposal is include population with a higher prevalence of lesions: individuals with positive FIT (fecal immunochemical test) in which the prevalence of lesions is 60%. In this case, sample size is reduced considerably.

The eligible population will be men and women, 50-69 years old, with no known risk factors and positive FIT.

Exclusion Criteria:

1. Individuals who have symptoms suggestive of colorectal disease (rectorrhagia, change in bowel movement frequency, constitutional syndrome, anaemia).
2. History of inflammatory bowel disease, colorectal polyposis, colorectal adenoma or CRC, and total or partial colectomy.
3. History of familial adenomatous polyposis or other hereditary polyposis syndromes; hereditary colorectal cancer not associated with polyposis (diagnosed by the presence of germinal mutation in the DNA repair genes and/or by fulfilment of the Amsterdam II criteria);
4. Severe co-morbidity that carries a poor short-term prognosis (disease with an average life expectancy of less than 5 years) or a chronic illness that involves significant limitation of physical activity.
5. Contraindication to undergoing colon capsule or virtual colonoscopy.

Study groups and randomisation:

All patients recruited who meet the inclusion criteria will be randomised into the two study groups:

Group I: Screening via virtual colonoscopy and subsequent conventional colonoscopy (within 1 week). In this group of patients, performance of the conventional colonoscopy will be delayed to ensure that bowel preparation is comparable in the two study groups.

Group II: Screening with colon capsule and subsequent conventional colonoscopy (within hours, since these patients will have already completed bowel preparation for the first screening test).

When the conventional colonoscopy is done, pertinent therapeutic procedures will be performed, if necessary.

Subsequently, the two groups of patients will be followed through visits to the hospital in which they will be instructed about the approach to follow from that time.

Sample size When we calculate the sample size we observed that we need more than 1000 patients per group. In this moment this study is very expensive and it is not feasible. Our proposal is include population with a higher prevalence of lesions: individuals with positive FIT (fecal immunochemical test) in which the prevalence of lesions is 60%. In this case, sample size is reduced considerably.

Adenomas detection rate (ADR) in these patients with positive FIT in colonoscopy (gold standard) is 60% (NEJM 2012). We assume that colon capsule will detect the same number of lesions than gold standard, and a difference of 15% with virtual colonoscopy will be clinically significant. We will need 187 patients per group, with a significance level of 5% and a statistical power of 80%.

The calculation was performed using the Study Size Granmo program.

ELIGIBILITY:
Inclusion Criteria:

The main objective in this study is compare two non-invasive techniques in the study of colorectal cancer. When we calculate the sample size we observed that we need more than 1000 patients per group. In this moment this study is very expensive and it is not feasible. Our proposal is include population with a higher prevalence of lesions: individuals with positive FIT (fecal immunochemical test) in which the prevalence of lesions is 60%. In this case, sample size is reduced considerably.

The eligible population will be men and women, 50-69 years old, with no known risk factors and positive FIT.

Exclusion Criteria:

1. Individuals who have symptoms suggestive of colorectal disease (rectorrhagia, change in bowel movement frequency, constitutional syndrome, anaemia).
2. History of inflammatory bowel disease, colorectal polyposis, colorectal adenoma or CRC, and total or partial colectomy.
3. History of familial adenomatous polyposis or other hereditary polyposis syndromes; hereditary colorectal cancer not associated with polyposis (diagnosed by the presence of germinal mutation in the DNA repair genes and/or by fulfilment of the Amsterdam II criteria);
4. Severe co-morbidity that carries a poor short-term prognosis (disease with an average life expectancy of less than 5 years) or a chronic illness that involves significant limitation of physical activity.
5. Contraindication to undergoing colon capsule or virtual colonoscopy.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population we are concerned with in this study is the healthy population-men and women 50-69 years of age with no significant history. Therefore, the screening method we offer must be the least invasive and the most comfortable method possible so that good compliance is achieved. This means techniques that are painless and essentially harmless in comparison with conventional colonoscopy. If we were to observe higher concordance between these techniques and conventional colonoscopy in terms of detecting lesions, we would use the latter strictly for therapeutic reasons in this population, thereby significantly reducing the complications associated with it
Sampling Method: Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with colorectal neoplastic lesions detected by colon capsule adn CTC | 3 years
  The primary endpoint was to compare the performance characteristics of CCE and CTC in detecting patients with colorectal neoplastic lesions, using colonoscopy as gold standard.

SECONDARY OUTCOMES:
number of advanced polypoid lesions and colorectal cancer (CRC) detected by CCE and CTC | 3 years
  (1) To compare the diagnostic rate of CCE and CTC in the detection of advanced colorectal neoplasms (i.e. advanced adenomas and CRC) using a threshold of >6 mm in size of lesions detected by any of these examinations to indicate the work-up colonoscopy.
Number of complications associated with each of the screening strategies | 3 years
  (2) To determine the incidence of adverse events (AE) associated with each screening strategy
Rate of false positives and false negatives obtained with CTC and colon capsule | 3 years
  (3) To determine the false-positive and false-negative rates of CCE and CTC in detecting significant colorectal neoplastic lesions as compared to colonoscopy.
Number of false negative lesions detected by CTC or colon capsule | 3 years
  (4) To determine significant independent predictive factors for false negative results in CTC or CCE

CONTACTS AND LOCATIONS:
Overall Officials: Begoña Gonzalez Suarez, PhMD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Spain

REFERENCES:
- [Derived] Gonzalez-Suarez B, Pages M, Araujo IK, Romero C, Rodriguez de Miguel C, Ayuso JR, Pozo A, Vila-Casadesus M, Serradesanferm A, Gines A, Fernandez-Esparrach G, Pellise M, Lopez-Ceron M, Flores D, Cordova H, Sendino O, Grau J, Llach J, Serra-Burriel M, Cardenas A, Balaguer F, Castells A. Colon capsule endoscopy versus CT colonography in FIT-positive colorectal cancer screening subjects: a prospective randomised trial-the VICOCA study. BMC Med. 2020 Sep 18;18(1):255. doi: 10.1186/s12916-020-01717-4. PMID 32943059